CLINICAL TRIAL: NCT00764725
Title: A Prospective Randomized, Open, Multi-Center Trial Comparing TNF-Blockade + MTX to MTX+SSZ+HCQ in Patients With Early RA With an Inadequate Response to MTX
Brief Title: Comparison of MTX+Anti-TNF to MTX+Conventional DMARDs in Patients With Early Rheumatoid Arthritis (RA) Who Failed MTX Alone (SWEFOT)
Acronym: SWEFOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Dr. Johan Bratt, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P0 3013 Swefot
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): MTX+SSZ+Plaquenil
  Interventions: Drug: conventional DMARD combination
- B (Active Comparator): MTX+Infliximab
  Interventions: Biological: MTX plus anti-TNF

INTERVENTIONS:
Drug: conventional DMARD combination — MTX+SSZ+Plaquenil; can be changed to MTX+cyclosporin within protocol
  Other Names: MTX=Methotrexate, SSZ=Sulfasalazine, Plaquenil=HCQ
  Arms: A
Biological: MTX plus anti-TNF — MTX + infliximab; can be changed to MTX + etanercept within protocol
  Other Names: infliximab=Remicade
  Arms: B

SUMMARY:
The Swefot trial was designed to compare two treatment strategies for patients with early rheumatoid arthritis (less than 1 year symptom duration): the use of a combination of traditional antirheumatic medications (DMARDs), versus a combination including a newer "biological" anti-TNF medication. In order to make this trial consistent with current practices in rheumatology, all patients were first given the most commonly used antirheumatic medication, methotrexate (MTX). After 3-4 months those patients who had not responded adequately to this treatment were randomized to receive either MTX plus sulfasalazine plus hydroxychloroquine, or MTX plus infliximab. Again, to be truly life-like, the trial allowed patients who could not tolerate one of the added medications to switch in treatment - but keeping with the same strategy - so that sulfasalazine plus hydroxychloroquine could be replaced by cyclosporin A, and infliximab by etanercept. The primary outcome in this trial was the percentage of patients who, after one year of treatment, achieved a "good response" as defined by Eular.

DETAILED DESCRIPTION:
The Swefot trial was designed to compare two treatment strategies for patients with early rheumatoid arthritis (less than 1 year symptom duration): the use of a combination of traditional antirheumatic medications (DMARDs), versus a combination including a newer "biological" anti-TNF medication. In order to make this trial consistent with current practices in rheumatology, all patients were first given the most commonly used antirheumatic medication, methotrexate (MTX). After 3-4 months those patients who had not responded adequately to this treatment were randomized to receive either MTX plus sulfasalazine plus hydroxychloroquine, or MTX plus infliximab. Again, to be truly life-like, the trial allowed patients who could not tolerate one of the added medications to switch in treatment - but keeping with the same strategy - so that sulfasalazine plus hydroxychloroquine could be replaced by cyclosporin A, and infliximab by etanercept. The primary outcome in this trial was the percentage of patients who, after one year of treatment, achieved a "good response" as defined by Eular. Secondary outcomes include Eular and ACR responses, HAQ and other QOL assessments, radiographic outcomes, and health-economic outcomes including EQ5D.

ELIGIBILITY:
Inclusion Criteria:

* RA, symptom duration < 12 months

Exclusion Criteria:

* Contraindication to any of the trial medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2002-12; Primary Completion 2007-04 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
EULAR individual response | 12 months

SECONDARY OUTCOMES:
All core set variables; function; x-ray; health-economic | 6-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Johan Bratt, MD PhD, Principal Investigator — Karolinska University Hospital

REFERENCES:
- [Derived] Miller H, Wallman JK, Petersson IF, Saevarsdottir S, Soderling J, Ernestam S, Askling J, van Vollenhoven R, Neovius M. Mortality over 14 years in MTX-refractory patients randomized to a strategy of addition of infliximab or sulfasalazine and hydroxychloroquine. Rheumatology (Oxford). 2021 May 14;60(5):2217-2222. doi: 10.1093/rheumatology/keaa553. PMID 33179071
- [Derived] Olofsson T, Wallman JK, Joud A, Schelin MEC, Ernestam S, van Vollenhoven R, Saevarsdottir S, Lampa J. Pain Over Two Years After Start of Biologic Versus Conventional Combination Treatment in Early Rheumatoid Arthritis: Results From a Swedish Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2021 Sep;73(9):1312-1321. doi: 10.1002/acr.24264. Epub 2021 Aug 2. PMID 32433827
- [Derived] Hambardzumyan K, Hermanrud C, Marits P, Vivar N, Ernestam S, Wallman JK, van Vollenhoven RF, Fogdell-Hahn A, Saevarsdottir S; SWEFOT study group. Association of female sex and positive rheumatoid factor with low serum infliximab and anti-drug antibodies, related to treatment failure in early rheumatoid arthritis: results from the SWEFOT trial population. Scand J Rheumatol. 2019 Sep;48(5):362-366. doi: 10.1080/03009742.2019.1602670. Epub 2019 Jun 27. PMID 31244356
- [Derived] Hambardzumyan K, Bolce RJ, Wallman JK, van Vollenhoven RF, Saevarsdottir S. Serum Biomarkers for Prediction of Response to Methotrexate Monotherapy in Early Rheumatoid Arthritis: Results from the SWEFOT Trial. J Rheumatol. 2019 Jun;46(6):555-563. doi: 10.3899/jrheum.180537. Epub 2019 Feb 1. PMID 30709958
- [Derived] Levitsky A, Brismar K, Hafstrom I, Hambardzumyan K, Lourdudoss C, van Vollenhoven RF, Saevarsdottir S. Obesity is a strong predictor of worse clinical outcomes and treatment responses in early rheumatoid arthritis: results from the SWEFOT trial. RMD Open. 2017 Aug 9;3(2):e000458. doi: 10.1136/rmdopen-2017-000458. eCollection 2017. PMID 28879052
- [Derived] Platten M, Kisten Y, Kalvesten J, Arnaud L, Forslind K, van Vollenhoven R. Fully automated joint space width measurement and digital X-ray radiogrammetry in early RA. RMD Open. 2017 Jun 29;3(1):e000369. doi: 10.1136/rmdopen-2016-000369. eCollection 2017. PMID 28879043
- [Derived] Hambardzumyan K, Saevarsdottir S, Forslind K, Petersson IF, Wallman JK, Ernestam S, Bolce RJ, van Vollenhoven RF. A Multi-Biomarker Disease Activity Score and the Choice of Second-Line Therapy in Early Rheumatoid Arthritis After Methotrexate Failure. Arthritis Rheumatol. 2017 May;69(5):953-963. doi: 10.1002/art.40019. Epub 2017 Mar 31. PMID 27992691
- [Derived] Eriksson JK, Wallman JK, Miller H, Petersson IF, Ernestam S, Vivar N, van Vollenhoven RF, Neovius M. Infliximab Versus Conventional Combination Treatment and Seven-Year Work Loss in Early Rheumatoid Arthritis: Results of a Randomized Swedish Trial. Arthritis Care Res (Hoboken). 2016 Dec;68(12):1758-1766. doi: 10.1002/acr.22899. PMID 27015295
- [Derived] Hambardzumyan K, Bolce RJ, Saevarsdottir S, Forslind K, Wallman JK, Cruickshank SE, Sasso EH, Chernoff D, van Vollenhoven RF. Association of a multibiomarker disease activity score at multiple time-points with radiographic progression in rheumatoid arthritis: results from the SWEFOT trial. RMD Open. 2016 Mar 1;2(1):e000197. doi: 10.1136/rmdopen-2015-000197. eCollection 2016. PMID 26958364
- [Derived] Levitsky A, Erlandsson MC, van Vollenhoven RF, Bokarewa MI. Serum survivin predicts responses to treatment in active rheumatoid arthritis: a post hoc analysis from the SWEFOT trial. BMC Med. 2015 Sep 30;13:247. doi: 10.1186/s12916-015-0485-2. PMID 26420684
- [Derived] van Vollenhoven RF, Bolce R, Hambardzumyan K, Saevarsdottir S, Forslind K, Petersson IF, Sasso EH, Hwang CC, Segurado OG, Geborek P. Brief report: enhancement of patient recruitment in rheumatoid arthritis clinical trials using a multi-biomarker disease activity score as an inclusion criterion. Arthritis Rheumatol. 2015 Nov;67(11):2855-60. doi: 10.1002/art.39274. PMID 26213309
- [Derived] Kastbom A, Forslind K, Ernestam S, Geborek P, Karlsson JA, Petersson IF, Saevarsdottir S, Klareskog L, van Vollenhoven RF, Lundberg K. Changes in the anticitrullinated peptide antibody response in relation to therapeutic outcome in early rheumatoid arthritis: results from the SWEFOT trial. Ann Rheum Dis. 2016 Feb;75(2):356-61. doi: 10.1136/annrheumdis-2014-205698. Epub 2014 Dec 30. PMID 25550338
- [Derived] Hambardzumyan K, Bolce R, Saevarsdottir S, Cruickshank SE, Sasso EH, Chernoff D, Forslind K, Petersson IF, Geborek P, van Vollenhoven RF. Pretreatment multi-biomarker disease activity score and radiographic progression in early RA: results from the SWEFOT trial. Ann Rheum Dis. 2015 Jun;74(6):1102-9. doi: 10.1136/annrheumdis-2013-204986. Epub 2014 May 8. PMID 24812287
- [Derived] Eriksson JK, Karlsson JA, Bratt J, Petersson IF, van Vollenhoven RF, Ernestam S, Geborek P, Neovius M. Cost-effectiveness of infliximab versus conventional combination treatment in methotrexate-refractory early rheumatoid arthritis: 2-year results of the register-enriched randomised controlled SWEFOT trial. Ann Rheum Dis. 2015 Jun;74(6):1094-101. doi: 10.1136/annrheumdis-2013-205060. Epub 2014 Apr 15. PMID 24737786
- [Derived] Saevarsdottir S, Rezaei H, Geborek P, Petersson I, Ernestam S, Albertsson K, Forslind K, van Vollenhoven RF; SWEFOT study group. Current smoking status is a strong predictor of radiographic progression in early rheumatoid arthritis: results from the SWEFOT trial. Ann Rheum Dis. 2015 Aug;74(8):1509-14. doi: 10.1136/annrheumdis-2013-204601. Epub 2014 Apr 4. PMID 24706006
- [Derived] Eriksson JK, Neovius M, Bratt J, Petersson IF, van Vollenhoven RF, Geborek P, Ernestam S. Biological vs. conventional combination treatment and work loss in early rheumatoid arthritis: a randomized trial. JAMA Intern Med. 2013 Aug 12;173(15):1407-14. doi: 10.1001/jamainternmed.2013.7801. PMID 23817631
- [Derived] van Vollenhoven RF, Geborek P, Forslind K, Albertsson K, Ernestam S, Petersson IF, Chatzidionysiou K, Bratt J; Swefot study group. Conventional combination treatment versus biological treatment in methotrexate-refractory early rheumatoid arthritis: 2 year follow-up of the randomised, non-blinded, parallel-group Swefot trial. Lancet. 2012 May 5;379(9827):1712-20. doi: 10.1016/S0140-6736(12)60027-0. Epub 2012 Mar 29. PMID 22464340
- [Derived] Saevarsdottir S, Wallin H, Seddighzadeh M, Ernestam S, Geborek P, Petersson IF, Bratt J, van Vollenhoven RF; SWEFOT Trial Investigators Group. Predictors of response to methotrexate in early DMARD naive rheumatoid arthritis: results from the initial open-label phase of the SWEFOT trial. Ann Rheum Dis. 2011 Mar;70(3):469-75. doi: 10.1136/ard.2010.139212. Epub 2010 Dec 13. PMID 21149498